CLINICAL TRIAL: NCT01729624
Title: A Qualitative Study Using Interviews With Patients Who Have Anti-neutrophil Cytoplasm Antibody (ANCA) Associated Vasculitis, to Develop a Patient Reported Outcome (PRO) Measure
Brief Title: PRO Development for ANCA Associated Vasculitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: Rec No: 12/SW/0252
Record Dates: First submitted 2012-10-25; First posted 2012-11-20 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Wegener Granulomatosis; Microscopic Polyangiitis; Churg-Strauss Syndrome
Keywords: Wegener Granulomatosis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Antibodies, Antineutrophil Cytoplasmic
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A qualitative study using interviews with patients who have antineutrophil cytoplasm antibody (ANCA) associated vasculitis, to develop a patient reported outcome (PRO)measure

DETAILED DESCRIPTION:
Patients with antineutrophil cytoplasmic antibody (ANCA) associated vasculitis (AAV) have inflammation in the small blood vessels leading to involvement in different body areas, e.g., the kidneys, lungs and skin. Untreated, the risk of death is over 80%; with current treatment, patients often suffer from ongoing disease activity, damage or treatment side effects which have a negative impact on quality of life. Because patients with AAV can have a wide range of disease features, the investigators hypothesise that general patient reported outcome (PROs) measurements, may not be specific enough to describe the full impact on quality of life.

The main objective of this project is to start from patients' experiences to develop a disease specific PRO for patients with AAV. Patients diagnosed with AAV will be recruited through clinics or inpatients at the Oxford University Hospitals (OUH) National Health Service (NHS) Trust, or, if the patients have previously consented to be contacted about future studies, through the Diagnostic and Classification of Vasculitis (DCVAS) or The Characterisation and Determinants of Quality of Life in ANCA Associated Vasculitis (VasQoL) study databases. After informed consent is obtained, individual patient interviews will be conducted; these will last for approximately one hour and will be recorded and transcribed. Themes will be independently extracted and amalgamated by the researchers. Approximately 25 patients with different types of ANCAassociated vasculitis and varying disease duration will be interviewed until saturation, i.e., no new substantive themes emerge. These themes will then evolve into individual candidate questionnaire items. Candidate items will be piloted on approximately 25 different patients with AAV using questionnaires and interviews, until no further comments arise, to produce a final set of candidate questionnaire items. The duration of the study 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female
* Aged 18 years or above (no upper limit).
* Diagnosed with granulomatosis with polyangiitis- Wegeners (GPA), Churg Strauss Syndrome (CSS) or microscopic polyangiitis (MPA)and fulfil either Chapel Hill consensus conference definitions or American College of Rheumatology (ACR) classification criteria.

Exclusion Criteria:

* Unable or unwilling to give independent written informed consent
* Significant communication barrier e.g., inability to speak English
* Membership of the steering committee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ANCA-associated vasculitis seen at the Oxford University Hospitals NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
This is a qualitative research study based on semi-quantitive exploratory patient interviews and therefore it is not appropriate to define only one outcome measure. | No formal outcome measure therefore not applicable
  The principle research objective: The investigators are going to interview patients with anti-neutrophil cytoplasm antibody associated vasculitis, to develop and pilot questionnaire items for a patient reported outcome measure specifically for their disease.
  The secondary research objective is to describe the impact of ANCA-associated vasculitis on the quality of life of patients attending the Oxford University Hospitals NHS Trust, based on individual anonymised interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom